CLINICAL TRIAL: NCT06410287
Title: Feasibility of an Art-based Intervention to Address Clinician Stigma and Improve Care for Neonatal Opioid Withdrawal Syndrome
Brief Title: Testing an Arts-based Program to Reduce Nurse Stigma Towards Perinatal Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Clayton John Shuman, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00248695; R21DA055067 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Nurse's Role; Stigma, Social; Implicit Bias
MeSH Terms: conditions — Social Stigma; Bias, Implicit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Site 1 (Experimental): Participants from the hospital randomized to the experimental group will be first to receive an invitation to complete the web-based educational program. The program will be open for one month. Thirty days after a participant completes the program, they will be sent a link to a follow up survey (web-based). At 60 days, participants who completed the program and the first follow up survey will be randomized to complete a second follow up survey or participate in a 1:1 interview.
  Interventions: Other: ArtSpective
- Site 2 (Other): Participants from the hospital randomized to the control setting will receive an invitation to complete a survey that collects baseline data for the outcome (stigma toward perinatal substance use) and demographic information. After thirty days, participants will be invited to complete the web-based educational program. Thirty days after completion, they will receive a link to a web-based follow up survey.
  Interventions: Other: ArtSpective

INTERVENTIONS:
Other: ArtSpective — ArtSpective is an interactive, educational program that uses art and museum-based pedagogy. The intervention is delivered asynchronously using a web-based platform. Participants engage with artwork, watch short educational videos, and read short clinical vignettes. After completing the program, participants receive a certificate of completion.

SUMMARY:
The goal of this pilot clinical trial is to evaluate the feasibility and limited effectiveness of a digital, arts-based educational intervention addressing nurse stigma towards perinatal substance use. The main questions it aims to answer are:

* What is the the feasibility of delivering the training through an asynchronous, web-based platform?
* What is the limited effectiveness of the program on nurse stigma towards perinatal substance use?

Participants will access and complete the training, including completion of a perinatal substance use stigma scale at baseline, immediately post, and 1-2 months month later. Participants will also be invited to participate in an interview.

Researchers will compare the intervention and control groups to see if the training reduces nurse stigma towards perinatal substance use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Licensed as a registered nurse
* Works at least part time
* Works on a labor, postpartum, nursery, neonatal intensive care, or pediatric unit in one of the participating hospitals

Exclusion Criteria:

* Works as per diem or agency nurse
* Not employed by a participating hospital
* Not a perinatal/pediatric nurse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Nurse Stigma toward Perinatal Substance Use | Measured at baseline, immediately post intervention, 30 days post, and 60 days post
  Negative or stigmatizing attitudes and/or beliefs registered nurses have towards perinatal substance use; measured using the Modified Attitudes About Drug Use in Pregnancy Scale. Total scores range between 1 and 5, with scores closer to 1 associated with a more positive outcome.

SECONDARY OUTCOMES:
Acceptability | immediately post intervention
  The level of satisfaction participants have towards the intervention; measured using an adapted version of the Abbreviated Acceptability Rating Profile. Total scores range from 1 to 5 with scores closer to 5 representing a more positive outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - ProMedica Toledo Hospital, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared upon request.